CLINICAL TRIAL: NCT00689546
Title: Natural Course of Acute Icteric Viral Hepatitis in Type II Diabetes Mellitus Patients and Non-Diabetic Patients:A Pilot Cohort Study
Brief Title: Acute Viral Hepatitis and Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: S K Acharya, All India Institute of Medical Sciences
Other Study IDs: KKS-AVH-2008
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2007-01

CONDITIONS: Acute Viral Hepatitis; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- I/A: All cases of acute viral hepatitis irrespective of type (A, B, E) with underlying Type 2 diabetes mellitus
- I/B: Age and sex matched non- diabetic patients with acute viral hepatitis (irrespective of type) recruited from all the patients of acute viral hepatitis registered during the time period in which cases were recruited.
- II/A: All diabetic who have acute icteric viral hepatitis due to HEV infection
- II/B: Age and sex matched diabetic who have acute icteric viral hepatitis due to hepatiits virus other than HEV.

SUMMARY:
It has been observed that several of patients having prolonged or complicated course of acute viral hepatitis have underlying diabetes. It is possible that with impaired hepatocyte regenerating capacity, these patients run a more prolonged and complicated course.

We hypothesize that acute hepatitis infection has a prolonged and complicated course among diabetic patients.

DETAILED DESCRIPTION:
Acute viral hepatitis is usually a self limited condition characterizes by typical course of prodrome followed by an icteric phase. In some cases the course may be protracted or complicated by the development of cholestatic phase or acute liver failure . The development of complicated course depends on a number of factors such as the type of virus and a variety of host factors including age of infection, immune status of the host and condition of the underlying liver before the onset of hepatitis.

Patients who have an underlying chronic liver disease or cirrhosis have increased risk of development of decompensation and liver related death when they develop superinfection with some hepatotropic viruses.

Vento etal demonstrated in their classical study that superinfection with hepatitis A on chronic liver disease is associated with high risk of decompensation and death. In India, since most of the adult population including those with chronic liver disease has been shown to have protective antibodies against HAV, this infection is rarely a problem in them.

Hepatitis E virus (HEV) has demonstrated to be the most common cause of acute hepatitis, acute liver failure and subacute liver in India. There is now enough data to suggest that HEV superinfection is also the commonest cause of acute decompensation of chronic liver disease in Indian subcontinent.

Many of these patients do not have any signs and symptoms of preexisting liver disease and it is the liver failure secondary to HEV superinfection which bring to light the underlying chronic liver disease.

World over, as well as in developing countries nonalcoholic fatty liver disease (NAFLD) is fast emerging as an important causes of chronic liver disease. Obesity and diabetes are two most important risk factors for NAFLD.It has been estimated that there would be about 366 million diabetes in the world by 2030.Of these 79.4 million will be in India.

Diabetes has been proposed as a risk factor for both chronic liver disease and HCC.The spectrum of liver involvement ranges from fatty liver, steatohepatitis, and fibrosis to cirrhosis. Even among patients with NASH, presence of diabetes is annotated with advanced stage of fibrosis . There is some suggestion that diabetic patients who develop acute viral hepatitis may have a prolonged course. Liver regeneration capacity has been demonstrated to be impaired among animal and human with fatty liver after partial resection. It is therefore possible that diabetic by of having NAFLD may have poor regenerating capacity leading to prolonged course of hepatitis.

It has been an observation in our unit that most of the patients who present with acute on chronic liver failure or subacute hepatic failure have diabetes. Whether it is simply a co-existence of two commonly occurring diseases (diabetes with a prevalence of 10% in Indian population and hepatitis E which is endemic(1) in our country) or the presence of acute hepatitis E in a diabetic patients some how produces a worse outcome as compared to hepatitis E in a non-diabetic patients. There fore it is important to find out the natural course of the two commonly occurring diseases when they occur together or separately.

We hypothesize that acute hepatitis infection has a prolonged and complicated course among diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 18 to 70 years

Exclusion Criteria:

* Recent intake of drugs known to cause acute hepatitis
* History of alcohol ingestion >40mg/day
* Suspected ischemic hepatitis
* Illness causing acute hepatitis such as Malaria hepatits, enteric hepatitis, Leptospirosis, septecemia
* HIV.
* Associated co morbidities, which can affect survival such as cardiovascular disease and diabetic nephropathy.
* Recent intake of drugs known to cause acute hepatitis
* History of alcohol ingestion >40mg/day
* Suspected ischemic hepatitis
* Malaria hepatits, enteric hepatitis, Leptospirosis, septecemia
* Co infection with HIV.
* Comorbidities which affect survival such as CAD and diabetic nephropathy.
* Gestational diabetes
* Pregnant female
* Cirrhosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients of acute viral hepatitis attending the OPD of Department of Gastroenterology and Endocrinology, All India Institute of Medical Sciences (AIIMS) will be candidates for the inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Duration of icteric hepatitis.

SECONDARY OUTCOMES:
Development of complications
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Subrat Acharya, DM, Principal Investigator — All India Institiute Of Medical Sciences
Locations (1):
- All India Institute Of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Hamid SS, Atiq M, Shehzad F, Yasmeen A, Nissa T, Salam A, Siddiqui A, Jafri W. Hepatitis E virus superinfection in patients with chronic liver disease. Hepatology. 2002 Aug;36(2):474-8. doi: 10.1053/jhep.2002.34856. PMID 12143058
- [Background] Monga R, Garg S, Tyagi P, Kumar N. Superimposed acute hepatitis E infection in patients with chronic liver disease. Indian J Gastroenterol. 2004 Mar-Apr;23(2):50-2. PMID 15176535
- [Background] Ramachandran J, Eapen CE, Kang G, Abraham P, Hubert DD, Kurian G, Hephzibah J, Mukhopadhya A, Chandy GM. Hepatitis E superinfection produces severe decompensation in patients with chronic liver disease. J Gastroenterol Hepatol. 2004 Feb;19(2):134-8. doi: 10.1111/j.1440-1746.2004.03188.x. PMID 14731121
- [Background] Vento S, Garofano T, Renzini C, Cainelli F, Casali F, Ghironzi G, Ferraro T, Concia E. Fulminant hepatitis associated with hepatitis A virus superinfection in patients with chronic hepatitis C. N Engl J Med. 1998 Jan 29;338(5):286-90. doi: 10.1056/NEJM199801293380503. PMID 9445408
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Behrns KE, Tsiotos GG, DeSouza NF, Krishna MK, Ludwig J, Nagorney DM. Hepatic steatosis as a potential risk factor for major hepatic resection. J Gastrointest Surg. 1998 May-Jun;2(3):292-8. doi: 10.1016/s1091-255x(98)80025-5. PMID 9841987